CLINICAL TRIAL: NCT05764252
Title: Utility of a Computational Biomarker (BioEP) in Supporting Clinicians' Decision Making in Patients Presenting to an Adult Epilepsy Service First-seizure Clinic: A Prospective Diagnostic Belief Updating Study.
Brief Title: A Prospective Diagnostic Belief Updating Study to verIfy the Utility of BioEP in First Seizure Clinics.
Acronym: PRISTINE
Status: Active, not recruiting | Type: Observational
Sponsor: Neuronostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NNBioEP001
Record Dates: First submitted 2023-02-15; First posted 2023-03-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; EEG; Biomarkers; diagnostic belief updating study; consultant nurse for the epilepsies; first seizure clinic; BioEP
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BioEP: The EEG will be analysed using the BioEP algorithm
  Interventions: Device: BioEP

INTERVENTIONS:
Device: BioEP — All patient's EEG will have the BioEP score conducted on it

SUMMARY:
The goal of this belief updating study is to assess the utility of BioEP as a complementary support tool in aiding clinical decision making in adults in first seizure clinics. The main outcomes we shall measure are:

* Clinicians' perception of seizure probability.
* Clinicians' decision to recommend commencing or deferring ASM (anti-seizure medications)
* Clinicians' decision to refer for additional investigations/services.

Participants will consent to have their EEG (that is taken at their routine care) to be used in the study. There is not extra burden to the participants taking part in the study.

DETAILED DESCRIPTION:
The accurate diagnosis and prognosis of epilepsy represents a significant unmet medical need. Due to the unpredictable nature of seizures, epilepsy is difficult to diagnose and treat. In the United Kingdom (UK), 125,000 people per annum are referred to first seizure clinics with suspected epilepsy of which 40,000 receive a confirmed diagnosis of epilepsy. Although diagnosing a patient with epilepsy is a clinical decision, clinicians often look towards diagnostic tests (such as electroencephalograms - EEGs) to support their decision-making process. At present, in the absence of observable epileptiform abnormalities (abnormal wave forms strongly associated with epilepsy on EEG, there are no clinically robust markers of epilepsy. Mathematical models provide a powerful and useful tool with which to identify and understand biological mechanisms that may lead to the risk of having seizures. By combining mathematical and computational techniques, Neuronostics have developed a biomarker called BioEP. Using properties in the background and clinically non contributary EEG, the investigators have demonstrated in retrospective, multi-site phase I and phase II studies sufficient evidence that could support clinicians to make more informed diagnostic decisions that investigators hope will lead to better and faster decisions about patients' diagnosis and treatment. The investigators will now conduct a prospective single site diagnostic belief updating study to examine the utility of BioEP in supporting clinicians' decision making a clinical setting in the NHS. The investigators will do this by inviting adults to take part who are suspected of having a first seizure and who will attend a first seizure clinic run by a Consultant Nurse for the Epilepsies (CNE) at the Royal Wolverhampton NHS trust. As part of the patients diagnostic work up, patients will have an EEG performed, the investigators will then apply BioEP to the patients EEG to derive a "risk score". This risk score will be presented to the CNE, who may then decide to combine it with the clinical history and clinical test information to help the CNE make decisions about patients' diagnosis and treatment.

The CNE will first rate the probability that the patient has experienced an epileptic seizure and probability of recurrence based on the clinical history and standard EEG (and any other standard tests ordered). A second assessment of this probability will be made after the CNE subsequently receives the BioEP risk score and report to quantify the updating of belief (that the patient has an increased seizure risk) and assess the utility of BioEP as a diagnostic decision support tool.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and above) presenting with first suspected seizure(s)
* Able to give informed consent
* Patient receives EEG following clinicians' decision to refer for an EEG based on clinical history and seizure description taken during first seizure clinic.

Exclusion Criteria:

* Participants unable to tolerate an EEG test so no EEG data was gathered
* Participants with a known hepatic/renal encephalopathy
* Participants that upon history taking have a clear clinical diagnosis of a physical condition other than epilepsy (e.g., vasovagal syncope)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (age 18 and above) presenting with first suspected seizure(s).
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Clinicians' perception of seizure probability in a 2 step process, using a 7-category scale and a 100-mm visual analogue scale | 1 day
  The clinician rates the probability that the patient will experience another epileptic seizure before and after the presentation of the BioEP score (updating beliefs). Using the clinician's ratings, we will impute the implicit individual likelihood ratios - the factor changes in the perceived odds of the patient experiencing another epileptic seizure based on the updated beliefs in the face of new evidence (the BioEP score)
Number of additional patient's investigations/services | 1 year
  Clinicians' decision-making over time will be explored. When patients present multiple times over a period, more clinical information is gathered and thus clinicians' perception of the probability of a seizure may change as evidence increases. The influence of multiple presentations and investigations shall be considered and reported descriptively. Any additional EEGs performed in the 1-year follow up period shall be analysed by our methods. The risk score will be presented to the CNE, who may then decide to combine it with any new emerging clinical history and clinical test information to help the CNE make any further decisions about patients' diagnosis and treatment.
Number of Clinicians' decisions to recommend commencing or deferring anti-seizure medications (ASM) | 1 year
  Clinicians' decision-making over time will be explored. The decisions to recommend commencing or deferring ASMs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Milaana Mainstone, Study Director — Neuronostics Ltd
Locations (1):
- Phil Tittensor, Wolverhampton, United Kingdom